CLINICAL TRIAL: NCT07179328
Title: Assessment of Safety and Feasibility of Focused Ultrasound Next Generational Dome Helmet Mediated Blood-Brain Barrier Disruption for the Treatment of High-Grade Glioma in Patients Undergoing Standard Chemotherapy
Brief Title: Focused Ultrasound Blood-Brain Barrier Disruption for the Treatment of High-Grade Glioma in Patients Undergoing Standard Chemotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB-6232
Record Dates: First submitted 2025-08-13; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: GBM; Glioblastoma Multiforme (GBM); Glioblastoma Multiforme of Brain; Glioblastoma Multiforme Glioma; HGG; Glioma; Brain Tumor Adult; Brain Tumor, Primary
Keywords: Focused Ultrasound; FUS; GBM; TMZ; Temozolomide; blood-brain barrier disruption (BBBD); MR-guided Focused Ultrasound (MRgFUS); Glioblastoma multiforme; blood-brain barrier opening; Drug delivery; Chemotherapy delivery
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focused Ultrasound BBB Disruption Using the Next Generation Dome Helmet and Definity (Experimental): Participants in this single-arm study will undergo repeated sessions (up to 6 cycles spaced 4-6 weeks apart) of focused ultrasound (FUS)-mediated blood-brain barrier (BBB) disruption using the Next Generation Dome Helmet (NGDH) during the maintenance phase of standard-of-care temozolomide (TMZ) chemotherapy. At the time of each FUS session, participants will receive their prescribed standard of care TMZ dose, as well as an intravenous injection of DEFINITY® ultrasound contrast agent that enables targeted BBB opening. Each session will be guided by MRI, and imaging will be used to assess the extent of BBB disruption. Clinical and safety assessments, blood sampling for biomarker analysis, and follow-up imaging will be conducted throughout the study period.
  Interventions: Device: Focused Ultrasound Next Generation Dome Helmet; Drug: Definity® Vial for (Perflutren Lipid Microsphere) Injectable Suspension

INTERVENTIONS:
Device: Focused Ultrasound Next Generation Dome Helmet — The Next Generation Dome Helmet (FUS NG) is a non-invasive, MRI-guided focused ultrasound system developed at Sunnybrook Research Institute. It is used to disrupt the blood-brain barrier (BBB) in patients with glioblastoma during the maintenance phase of temozolomide (TMZ) therapy. The device allows targeted BBB opening using a fixed transducer array and intravenous DEFINITY® contrast.
Drug: Definity® Vial for (Perflutren Lipid Microsphere) Injectable Suspension — DEFINITY® Perflutren Injectable Microbubbles is an ultrasound contrast imaging agent that will be used for blood brain barrier opening during focused ultrasound. These microbubbles will be injected during the focused ultrasound procedure.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and feasibility of focused ultrasound (FUS)-mediated blood-brain barrier (BBB) disruption using the Next Generation Dome Helmet (NGDH) in adults with glioblastoma (GBM) undergoing the maintenance phase of the standard "Stupp protocol".

Participants will:

* Undergo repeated FUS BBB disruption treatments during the maintenance phase of temozolomide (TMZ) chemotherapy.
* Receive intravenous ultrasound contrast (DEFINITY®) prior to each FUS session to facilitate targeted BBB disruption.
* Undergo serial MRI scans and clinical assessments to evaluate safety and the extent of BBB opening.
* Provide blood samples (and tumor tissue if available) for biomarker analysis related to BBB permeability, tumor presence, and treatment response.
* Be followed for progression-free survival (PFS) and overall survival (OS) during routine neuro-oncology visits until end of life.

DETAILED DESCRIPTION:
This is a Phase I, single-center, single-arm clinical trial. Approximately 10 participants are expected to be enrolled. The active therapy phase for participants will last approximately 6 to 8 months. Information about each participant's condition will continue to be collected for as long as possible to evaluate the effects of the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years, inclusive.
2. Able and willing to provide written informed consent.
3. Diagnosis of Glioblastoma by histology or molecular markers based on WHO 2021 classification.
4. Previously undergone a maximal safe surgical resection and completed concurrent, standard-of-care RT and TMZ without any complications and deemed eligible for the maintenance phase of TMZ treatment.
5. Tumor or tumor resection cavity is clearly defined on screening MRI scans.
6. Karnofsky Performance Score rating 70-100.
7. American Society of Anesthesiologists (ASA) physical status score of 1-3.
8. Life expectancy of at least 3 months and able to attend all study visits.

Exclusion Criteria:

1. Patients presenting with the following imaging characteristics:

   i. Following steroid treatment, brain edema and/or mass effect that causes midline shift or shift in wall of the third ventricle of more than 10 mm.

   ii. Evidence of recent (less than 2 weeks) intracranial hemorrhage. iii. Calcifications in the FUS sonication beam path in the event system tools cannot tailor the treatment around these calcification spots.
2. The sonication pathway to the tumor involves:

   i. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp.

   ii. Clips or other metallic implanted objects in the skull or the brain, except shunts.
3. The subject presents with symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, and papilledema).
4. Patients requiring increasing doses of corticosteroids.
5. Patient receiving bevacizumab (Avastin) therapy.
6. Patients with ≥25% increase in volume of contrast enhancement at time of assessment for study enrollment, compared with their first postoperative MRI. This cut-off is used to differentiate between pseudoprogression (which can occur following both radiation and TMZ therapy) and true tumor progression. This will be further ascertained through a discussion between the study neurosurgeons and radiologists.
7. Patients undergoing other concurrent therapies such as chemotherapy wafers, immunotoxins delivered by convection-enhanced delivery, regionally administered gene and viral therapies, immunotherapies, and focal irradiation with brachytherapy, stereotactic radiosurgery, and laser interstitial thermotherapy. These regimens have been shown to cause contrast enhancement in the resection cavity boundary, which can be difficult to differentiate from true tumor recurrence.
8. Cardiac disease or unstable hemodynamics including:

   i. Documented myocardial infarction within six months of enrollment. ii. Unstable angina on medication. iii. Congestive heart failure. iv. Left ventricular ejection fraction <50%. v. History of a hemodynamically unstable cardiac arrhythmia. vi. Cardiac pacemaker.
9. Severe hypertension (diastolic blood pressure (DBP) > 100 on medication).
10. Anti-coagulant therapy, or medications known to increase risk of hemorrhage within washout period prior to treatment (i.e., antiplatelet or vitamin K inhibitor anticoagulants within 7 days, non-vitamin K inhibitor anticoagulants within 72 hours, or heparin-derived compounds within 48 hours of treatment).
11. History of a bleeding disorder, coagulopathy or with a history of spontaneous tumor hemorrhage.
12. Abnormal level of platelets (< 100,000) or INR > 1.3.
13. Documented cerebral infarction within the past 12 months.
14. TIA in the last 1 month.
15. Cerebral or systemic vasculopathy.
16. Insulin-dependent diabetes mellitus that is not well-controlled or that in the Investigator's opinion precludes participation in the study.
17. Known sensitivity to gadolinium-DTPA.
18. Known sensitivity to DEFINITY® ultrasound contrast agent or perflutren.
19. Contraindications to MRI such as non-MRI-compatible implanted devices, unable to tolerate an MRI due to for instance pain or claustrophobia, untreated, uncontrolled sleep apnea.
20. Positive pregnancy test (for pre-menopausal women).
21. Known life-threatening systemic disease.
22. Severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 and/or on dialysis.
23. Right to left or bi-directional cardiac shunt.
24. Previous full course of chemotherapy for GBM (at the discretion of investigator).
25. Previous radiotherapy.
26. Allergy to eggs or egg products.
27. Subjects with evidence of cranial or systemic infection.
28. Subjects with chronic pulmonary disorders.
29. Subjects with a history of drug allergies, asthma or hay fever, and multiple allergies, in particular subjects with a history of anaphylaxis.
30. Subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation, or QT prolongation observed on screening ECG (QTc > 450 for men and >470 for women).
31. Subjects with evidence of Hepatitis B virus infection/carrier state.
32. Liver injury as indicated by liver function tests that in the Investigator's opinion precludes participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Safety of Focused Ultrasound-Mediated BBB Disruption | Participants will be evaluated at baseline, every 8 weeks during the first year, and every 12 weeks during the second year.
  Safety will be evaluated by monitoring the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) related to FUS BBB disruption, graded according to the Common Terminology Criteria for Adverse Events (CTCAE). Neurological assessments and MRI findings will be used to support safety evaluation.

SECONDARY OUTCOMES:
Clinical Efficacy - Radiographic Response (per modified RANO criteria) | Participants will be evaluated at baseline, every 8 weeks during the first year, and every 12 weeks during the second year.
  Tumor response will be evaluated using MRI imaging and assessed according to modified Response Assessment in Neuro-Oncology (RANO) criteria.
Clinical Efficacy - Progression-Free Survival and Overall Survival | Participants will be evaluated at baseline, every 8 weeks during the first year, and every 12 weeks during the second year.
  Comparing the PFS (by RANO 2.0 criteria) and Overall Survival (OS) of patients to historical controls.
Clinical Efficacy - Comparison of liquid and tumour tissue biomarkers in relation to BBB disruption. | Assessed at baseline and 1 day post-treatment for each of the 6 BBBD treatment cycles
  Blood samples will be analyzed for BBB disruption and tumour-related biomarkers, including S100β protein, inflammatory cytokines, circulating DNA, exosomes, and circulating tumour cells. The specific biomarkers analyzed will be determined by the investigator based on sample availability.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No